CLINICAL TRIAL: NCT00871715
Title: Interdisciplinary Comprehensive Arm Rehab Evaluation (ICARE) Stroke Initiative
Brief Title: Arm Rehabilitation Study After Stroke
Acronym: ICARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carolee Winstein, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01NS056256 (NIH); U01NS056256 (NIH)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Stroke; Brain Infarction; Brain Ischemia; Cerebral Infarction; Cerebrovascular Disorders
Keywords: stroke; hemiparesis; physical therapy; occupational therapy; neurorehabilitation; patient focused; motor learning; motor control; skill acquisition; skill training; motor recovery; task oriented training; task specific training; arm function; hand function; upper extremity; arm therapy; physical rehabilitation; arm rehabilitation; motor function
MeSH Terms: conditions — Stroke; Brain Infarction; Brain Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded to treatment allocation
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASAP (Experimental): A focused, intense, evidence-based, upper extremity rehabilitation program, administered during the early post-acute outpatient interval. The training intervention is based on the fundamental elements of skill acquisition through task-specific practice, impairment mitigation to increase capacity, and motivational enhancements to build self-confidence.
  Interventions: Behavioral: Accelerated Skill Acquisition Program (ASAP)
- DEUCC (Active Comparator): Dose-equivalent usual and customary arm therapy administered early post-acutely in the outpatient setting. This is a 30-hour dose equivalency group, administered over 1-hour visits at a frequency of 3x/week for a 10-week duration.
  Interventions: Behavioral: Dose-Equivalent Usual & Customary Care - DEUCC
- UCC (Other): Usual and customary arm therapy administered early post-acutely in the outpatient setting. This is an observation only group with treatment dose administered in accordance with usual and customary practices.
  Interventions: Behavioral: Usual and Customary Care - UCC

INTERVENTIONS:
Behavioral: Accelerated Skill Acquisition Program (ASAP) — A 30-hour dose is administered over 1-hour visits at a frequency of 3x/week for a 10-week duration. A 2-hour orientation/evaluation session precedes the first visit.
  Other Names: ASAP
  Arms: ASAP
Behavioral: Dose-Equivalent Usual & Customary Care - DEUCC — Usual and customary arm therapy administered early post-acutely in the outpatient setting, adjusted for dose, but otherwise administered in accordance with usual and customary practices. This is a 30-hour dose equivalency group, administered over 1-hour visits at a frequency of 3x/week for a 10-week duration.
  Other Names: DEUCC
  Arms: DEUCC
Behavioral: Usual and Customary Care - UCC — Usual and customary arm therapy administered early post-acutely in the outpatient setting. This is an observation only group and treatment dose will be administered in accordance with usual and customary practices.
  Other Names: UCC
  Arms: UCC

SUMMARY:
This study is about arm and hand recovery after a stroke. The investigators are testing an experimental arm therapy called Accelerated Skill Acquisition Program (ASAP) which combines challenging, intensive and meaningful practice of tasks of the participant's choice compared to two standard types of therapy (usual and customary arm therapy totaling 30 hours and usual and customary arm therapy for a duration indicated on the therapy prescription). A second objective is to characterize current outpatient arm therapy (dosage & content) following stroke for individuals who are eligible for ICARE. Eligible candidates must have had a stroke affecting an arm within the last 106 days.

DETAILED DESCRIPTION:
Of the 700,000 individuals who experience a new or recurrent stroke each year, a majority have considerable residual disability. Sixty-five percent (65%) of patients at 6 months are unable to incorporate the paretic hand effectively into daily activities. In turn, this degree of functional deficit contributes to a reduced quality of life after stroke. The extent of disability has been underplayed by the use of the Barthel Index that captures only basic activities of daily living such as self-care and does not extend to activities and participation at higher levels of functioning that are most affected by a residual upper extremity disability. The past decade has witnessed an explosion of different therapy interventions designed to capitalize on the brain's inherent capability to rewire and learn well into old age and more importantly for rehabilitation, after injury. The most effective arm-focused interventions with the strongest evidence and potentially the most immediate and cost-effective appeal for the current health-care environment share a common emphasis on focused task-specific training applied with an intensity higher than usual care. Therefore, our primary aim is to compare the efficacy of a fully defined, hybrid combination of the most effective interventions (forced-use/constraint-induced therapy and skill-based/impairment-mitigating motor learning training), the Accelerated Skill Acquisition Program (ASAP), to an equivalent dose of usual and customary outpatient therapy.

ELIGIBILITY:
INCLUSION

Ischemic or hemorrhagic stroke.

Hemiparesis in an upper extremity.

Age 21+.

Able to communicate in English (or Spanish,Rancho Los Amigos site only).

Willing to attend outpatient therapy & f/u evaluations for 1 yr.

Some active finger extension.

EXCLUSION

Traumatic or non-vascular brain injury, subarachnoid hemorrhage, AV malformation.

History of psychiatric illness requiring hospitalization within past 24 mos.

Active drug treatment for dementia.

Neurologic condition that may affect motor response (e.g. Parkinson's, ALS, MS).

History of head trauma requiring >48 hours of hospitalization within past 12 mos.

Amputation of all fingers or thumb of hemiparetic (weak) arm.

Treated with Botox in affected arm within last 3 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2009-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolee J. Winstein, PhD, PT, Principal Investigator — University of Southern California; Alexander Dromerick, MD, Principal Investigator — MedStar National Rehabilitation Network; Steven Wolf, PhD, PT, Principal Investigator — Emory University; Monica A Nelsen, DPT, PT, Study Director — University of Southern California
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Rancho Los Amigos National Rehabilitation Center, Los Angeles, California
  - Long Beach Memorial Medical Center, Los Angeles, California
  - Huntington Rehabilitation Medicine Associates, Los Angeles, California
  - Casa Colina Centers for Rehabilitation, Los Angeles, California
  - National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia

REFERENCES:
- [Background] Winstein CJ, Wolf SL, Dromerick AW, Lane CJ, Nelsen MA, Lewthwaite R, Blanton S, Scott C, Reiss A, Cen SY, Holley R, Azen SP; ICARE Investigative Team. Interdisciplinary Comprehensive Arm Rehabilitation Evaluation (ICARE): a randomized controlled trial protocol. BMC Neurol. 2013 Jan 11;13:5. doi: 10.1186/1471-2377-13-5. PMID 23311856
- [Background] Duff SV, He J, Nelsen MA, Lane CJ, Rowe VT, Wolf SL, Dromerick AW, Winstein CJ. Interrater reliability of the Wolf Motor Function Test-Functional Ability Scale: why it matters. Neurorehabil Neural Repair. 2015 Jun;29(5):436-43. doi: 10.1177/1545968314553030. Epub 2014 Oct 16. PMID 25323459
- [Result] Winstein CJ, Wolf SL, Dromerick AW, Lane CJ, Nelsen MA, Lewthwaite R, Cen SY, Azen SP; Interdisciplinary Comprehensive Arm Rehabilitation Evaluation (ICARE) Investigative Team. Effect of a Task-Oriented Rehabilitation Program on Upper Extremity Recovery Following Motor Stroke: The ICARE Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):571-81. doi: 10.1001/jama.2016.0276. PMID 26864411
- [Derived] Martinez C, Bacon H, Rowe V, Russak D, Fitzgerald E, Woodbury M, Wolf SL, Winstein C. A Reaching Performance Scale for 2 Wolf Motor Function Test Items. Arch Phys Med Rehabil. 2020 Nov;101(11):2015-2026. doi: 10.1016/j.apmr.2020.05.003. Epub 2020 May 17. PMID 32433993
- [Derived] Lewthwaite R, Winstein CJ, Lane CJ, Blanton S, Wagenheim BR, Nelsen MA, Dromerick AW, Wolf SL. Accelerating Stroke Recovery: Body Structures and Functions, Activities, Participation, and Quality of Life Outcomes From a Large Rehabilitation Trial. Neurorehabil Neural Repair. 2018 Feb;32(2):150-165. doi: 10.1177/1545968318760726. PMID 29554849
- [Derived] Rowe VT, Winstein CJ, Wolf SL, Woodbury ML. Functional Test of the Hemiparetic Upper Extremity: A Rasch Analysis With Theoretical Implications. Arch Phys Med Rehabil. 2017 Oct;98(10):1977-1983. doi: 10.1016/j.apmr.2017.03.021. Epub 2017 Apr 21. PMID 28434819
- See also: ICARE Administrative Headquarters: USC Department of Biokinesiology & Physical Therapy — http://pt.usc.edu/
- See also: ICARE Clinical Site: Casa Colina Rehabilitation Centers — http://www.casacolina.org/A-Center-of-Excellence/Signature-Programs/Stroke/Clinical-Trials.aspx
- See also: ICARE Clinical Center: National Rehabilitation Hospital — http://www.nrhrehab.org
- See also: ICARE Clinical Site: Huntington Rehabilitation Medical Associates — http://huntingtonrehab.com/
- See also: ICARE Clinical Site: Rancho Los Amigos National Rehabilitation Center — http://www.rancho.org
- See also: ICARE Clinical Center: Emory University — http://www.rehabmed.emory.edu
- See also: ICARE Clinical Site: Long Beach Memorial Medical Center — http://www.memorialcare.org/long_beach/about.cfm
- See also: ICARE Clinical Site: Cedars Sinai Medical Center — http://www.cedars-sinai.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 5 and 106 days post-stroke, predominantly during inpatient rehabilitation, from 7 sites in the United States metropolitan areas of Los Angeles, CA, Atlanta, GA and Washington, D.C.
Pre-assignment Details: From June 2009 through February 2013, 11,051 patients were pre-screened (medical record review) followed by 772 in-person screening assessments. Through both processes, 9,219 were excluded because they did not meet eligibility criteria; 645 declined and 826 were excluded for other reasons.
Groups:
- ASAP Accelerated Skill Acquisition Program: A structured, evidence-based, task-oriented rehabilitation program was administered during the early post-acute outpatient interval. It focused entirely on recovery of the affected upper extremity. The training intervention was based on the fundamental elements of skill acquisition through intense bouts of task-specific practice, impairment mitigation (strengthening exercises, shoulder stability/mobility, etc.) to increase capacity, and motivational enhancements to build self-confidence and autonomy.
  Accelerated Skill Acquisition Program (ASAP): The prescribed dose was 30-hours administered over 1-hour visits at a frequency of 3x/week for a 10-week duration. A 2-hour orientation/evaluation session preceded the first visit.
- DEUCC Dose-Equivalent Usual & Customary Care: Therapy content was not structured or standardized across therapists or sites. Usual and customary occupational therapy was adjusted for dose and administered early post-acutely in the outpatient setting. It consisted of usual and customary outpatient occupational therapy according to local practices, payer guidelines and participant preferences. It may have focused on more diverse needs than the affected upper extremity.
  Dose-Equivalent Usual & Customary Care (DEUCC): This group was prescribed a 30-hour dose equivalency, administered over 1-hour visits at a frequency of 3x/week for a 10-week duration.
- UCC Usual & Customary Care: Therapy content was not structured or standardized across therapists or sites. Usual and customary occupational therapy was administered early post-acutely in the outpatient setting according to local practices, payer guidelines and participant preferences. It may have focused on more diverse needs than the affected upper extremity.
  Usual and Customary Care (UCC): This was an observation only group; treatment dose was prescribed and provided in accordance with usual and customary practices.
Period: Overall Study
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Started | 119 | 120 | 122
Post-Intervention | 112 | 115 | 115
6-mo Follow-up | 110 | 113 | 112
Completed | 104 ("Completed" refers to participants who completed the primary outcome, Wolf Motor Function Test.) | 104 ("Completed" refers to participants who completed the primary outcome, Wolf Motor Function Test.) | 96 ("Completed" refers to participants who completed the primary outcome, Wolf Motor Function Test.)
Not Completed | 15 | 16 | 26
Not completed — Withdrawal by Subject | 6 | 10 | 15
Not completed — Physician Decision | 6 | 0 | 2
Not completed — Lost to Follow-up | 3 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care | Total
Number analyzed (Participants) | 119 | 120 | 122 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.7) | 59.9 (10.5) | 61.1 (13.1) | 60.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 50 | 158
  Male | 64 | 67 | 72 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-selected from categories determined in 1997 by the U.S. Office of Management and Budget in accordance with sponsor mandate.
  Participants
    Hispanic or Latino | 9 | 14 | 13 | 36
    Not Hispanic or Latino | 107 | 106 | 107 | 320
    Unknown or Not Reported | 3 | 0 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-selected from categories determined in 1997 by the U.S. Office of Management and Budget in accordance with sponsor mandate. For this self-selected measure, 35 participants (9 ASAP, 12 DEUCC, 14 UCC) specified other categories to identify their race. Since an "Other" field is not available, these 35 are included in the count under "Unknown or Not reported"
  Participants
    American Indian or Alaska Native | 4 | 1 | 0 | 5
    Asian | 9 | 7 | 3 | 19
    Native Hawaiian or Other Pacific Islander | 3 | 1 | 3 | 7
    Black or African American | 47 | 50 | 54 | 151
    White | 38 | 43 | 43 | 124
    More than one race | 3 | 3 | 1 | 7
    Unknown or Not Reported | 15 | 15 | 18 | 48
Region of Enrollment [Number; unit: participants]
  United States | 119 | 120 | 122 | 361
Education [Number; unit: participants] — Highest level of education completed (self-reported)
  participants
    Less than high school | 4 | 2 | 2 | 8
    Some high school | 6 | 12 | 8 | 26
    Completed high school | 24 | 21 | 27 | 72
    Some college | 42 | 42 | 46 | 130
    Completed bachelor's degree | 22 | 26 | 23 | 71
    Completed master's degree | 15 | 11 | 7 | 33
    Completed doctoral degree | 6 | 6 | 8 | 20
    Unknown or Not Reported | 0 | 0 | 1 | 1
Referral source [Number; unit: participants] — Setting in which participant was first prospectively identified.
  participants
    Inpatient rehabilitation | 80 | 79 | 88 | 247
    Outpatient | 6 | 5 | 5 | 16
    Acute care | 21 | 26 | 19 | 66
    Transitional day program | 3 | 2 | 2 | 7
    Open referral | 9 | 7 | 8 | 24
    Other | 0 | 1 | 0 | 1
Language [Number; unit: participants]
  English | 117 | 119 | 121 | 357
  Spanish | 2 | 1 | 1 | 4
Time from stroke to randomization [Mean (Standard Deviation); unit: days] | 45.2 (20.3) | 45.0 (22.8) | 47.0 (23.9) | 45.8 (22.4)
Stroke type [Number; unit: participants]
  Ischemic without hemorrhagic conversion | 100 | 98 | 101 | 299
  Ischemic with hemorrhagic conversion | 3 | 4 | 4 | 11
  Intraparenchymal hemorrhagic | 16 | 12 | 15 | 43
  Other | 0 | 5 | 1 | 6
  Unknown or Not Reported | 0 | 1 | 1 | 2
Stroke location [Number; unit: participants]
  Right hemisphere | 57 | 56 | 60 | 173
  Left hemisphere | 49 | 55 | 50 | 154
  Cerebellum | 0 | 1 | 0 | 1
  Brain stem | 11 | 5 | 9 | 25
  Other | 2 | 3 | 3 | 8
Side of hemiparesis [Number; unit: participants]
  Right | 51 | 60 | 57 | 168
  Left | 68 | 60 | 65 | 193
Stroke severity [Mean (Standard Deviation); unit: units on a scale] — Upper Extremity Motor Fugl Meyer total score range 0-66; eligible range: 19-58. A lower score indicates greater impairment. For stratification purposes: low severity is greater than or equal to 36; high severity is less than 36.
  National Institutes of Health Stroke Scale total score range 0-42; higher values represent greater severity.
  units on a scale
    Upper Extremity Motor Fugl-Meyer score | 41.7 (9.5) | 41.5 (9.2) | 41.6 (9.5) | 41.6 (9.4)
    National Institutes of Health Stroke Scale score | 3.6 (2.0) | 3.4 (1.7) | 3.7 (1.7) | 3.6 (1.8)
Strata [Number; unit: participants] — Severity: Upper extremity motor Fugl-Meyer score eligible range: 19-58 (low severity is greater than 35; high severity is less than 36).
  Stroke onset, time to randomization: eligible range: 14-106 days (early onset is less than 60 days; late onset is greater than 59 days).
  participants
    Low severity, early onset | 68 | 70 | 67 | 205
    Low severity, late onset | 16 | 16 | 18 | 50
    High severity, early onset | 23 | 22 | 25 | 70
    High severity, late onset | 12 | 12 | 12 | 36
Concordance [Number; unit: participants] — Concordant: the paretic limb is the dominant limb. Discordant: the paretic limb is the non-dominant limb.
  participants
    Concordant | 55 | 64 | 57 | 176
    Discordant | 64 | 56 | 65 | 185
Pre-randomization outpatient occupational therapy [Number; unit: participants] | 34 | 29 | 42 | 105
Amount of pre-randomization outpatient occupational therapy [Mean (Standard Deviation); unit: hours] | 4.4 (3.1) | 3.3 (2.3) | 3.7 (3.4) | 3.8 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test (WMFT) Log-transformed Time
Description: Change from baseline to end-of-study (12 months post-randomization) in log-transformed time required to perform each of the 15 standardized tasks with each upper extremity.
Time Frame: Baseline to 1 year post-randomization
Population: Number analyzed reflects actual evaluations completed, which varied by outcome assessment. All analyses were also performed in accord with the pre-planned intent-to-treat (ITT) principle with multiple imputation, comparing outcomes by assigned group. No differences were observed between imputed models and actual complete case data.
Measure: Mean (95% Confidence Interval); unit: log(seconds)
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 104 | 104 | 96
log(seconds) | -0.8 [-1.0 to -0.6] | -0.9 [-1.0 to -0.7] | -0.8 [-1.0 to -0.6]

2. Primary Outcome: Wolf Motor Function Test Time
Description: Change from baseline to end-of-study (12 months post-randomization) in time required to perform each of the 15 standardized tasks with each upper extremity.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 104 | 104 | 96
seconds | -8.1 [-11.7 to -4.5] | -8.7 [-11.6 to -5.8] | -7.5 [-10.5 to -4.6]

3. Primary Outcome: Stroke Impact Scale (SIS) Hand Function Subscale Score.
Description: Change from baseline to end-of-study (one year post-randomization). Range: 0-100; positive values reflect an improvement. Higher values indicate better perception of hand function.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 105 | 107 | 101
units on a scale | 37.6 [31.7 to 43.5] | 35.7 [30.4 to 40.9] | 37.1 [32.2 to 42.1]

4. Primary Outcome: Stroke Impact Scale (SIS), Hand Function Subscale, Percentage of Participants That Improved at Least 25 Points From Baseline to End-of-study (One Year Post-randomization)
Description: The available range for improvement is from 0-100; thus participants with a baseline SIS score greater than 75 (n=15) were excluded from these analyses.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 99 | 104 | 99
percentage of participants | 72.7 | 72.1 | 68.7

5. Secondary Outcome: Wolf Motor Function Test (WMFT) Functional Ability Scale (FAS)
Description: Assesses movement quality via digital media review of task performance post hoc, rated on a 6-point ordinal scale.
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

6. Secondary Outcome: Stroke Impact Scale (SIS) Mobility Subscale Score.
Description: Change from baseline to end-of-study (one year post-randomization). Range: 0-100; positive values reflect an improvement. Higher values indicate better perception of mobility.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 105 | 107 | 101
units on a scale | 11.22 (22.53) | 12.08 (21.15) | 14.91 (22.6)

7. Secondary Outcome: Stroke Impact Scale (SIS) ADL/IADL Subscale Score.
Description: Change from baseline to end-of-study (one year post-randomization). Range: 0-100; positive values reflect an improvement. Higher values indicate better perception of ease with activities queried.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 105 | 107 | 101
units on a scale | 22.69 (20.33) | 21.53 (18.76) | 23.22 (18.88)

8. Secondary Outcome: National Institute of Health Stroke Scale (NIHSS)
Description: Change from baseline to end-of-study (12 months post-randomization) in National Institute of Health Stroke Scale (NIHSS). Range 0-2. Lower scores indicate less stroke severity.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 104 | 104 | 91
score on a scale | -1.67 (2.28) | -1.61 (1.79) | -1.76 (1.7)

9. Secondary Outcome: Wolf Motor Function Test (WMFT) Strength Component, Task #7 Weight to Box
Description: Wolf Motor Function Test (WMFT) strength component, Task #7 Weight to Box, measured in pounds.
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

10. Secondary Outcome: Wolf Motor Function Test (WMFT) Strength Component, Task #14 Grip Strength
Description: Wolf Motor Function Test (WMFT) strength component, Task #14 Grip strength, measured in kilograms, change from baseline to one year post-randomization.
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

11. Secondary Outcome: Arm Muscle Torque Test - Elbow Extensors
Description: Change from baseline to end-of-study (12 months post-randomization) in isometric torque generated as measured in kilograms using a hand held Lafayette manual muscle test dynamometer and standard testing positions.Positive values indicate a strength gain.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 95 | 98 | 85
kilograms | 20.0 (47.33) | 15.73 (48.10) | 14.58 (50.28)

12. Secondary Outcome: Arm Muscle Torque Test - Elbow Flexors
Description: Change from baseline to end-of-study (12 months post-randomization) in isometric torque generated as measured in kilograms using a hand held Lafayette manual muscle test dynamometer and standard testing positions. Positive values indicate a strength gain.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 95 | 99 | 85
kilograms | 30.41 (52.03) | 20.78 (56.39) | 24.21 (45.13)

13. Secondary Outcome: Arm Muscle Torque Test - Shoulder Extensors
Description: as for outcome 12
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 91 | 94 | 79
kilograms | 25.61 (56.63) | 20.76 (55.23) | 18.64 (59.04)

14. Secondary Outcome: Arm Muscle Torque Test - Shoulder Flexors
Description: as for outcome 12
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 90 | 93 | 79
kilograms | 21.41 (57.12) | 24.4 (51.90) | 19.74 (47.86)

15. Secondary Outcome: Arm Muscle Torque Test - Wrist Extensors
Description: as for outcome 12
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 95 | 97 | 85
kilograms | 15.19 (37.59) | 18.07 (34.03) | 18.12 (32.07)

16. Secondary Outcome: Arm Muscle Torque Test - Wrist Flexors
Description: as for outcome 12
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 93 | 99 | 85
kilograms | 16.24 (39.37) | 10.71 (30.21) | 8.96 (28.76)

17. Secondary Outcome: As-Tex Sensory Index
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

18. Secondary Outcome: Upper Extremity Fugl Meyer (UEFM), Motor Component
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

19. Secondary Outcome: D-KEFS Verbal Fluency Test
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

20. Secondary Outcome: Digits Span Backward
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

21. Secondary Outcome: Hopkins Verbal Learning Test, Revised (HVLT-R)
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

22. Secondary Outcome: Color Trails Making Tests 1 & 2
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

23. Secondary Outcome: Short Blessed Memory Test
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

24. Secondary Outcome: Patient Health Questionnaire 9 (PHQ-9)
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

25. Secondary Outcome: Confidence in Arm & Hand Movement (CAHM)
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

26. Secondary Outcome: Stroke Impact Scale (SIS) Communication Subscale Score.
Description: Change from baseline to end-of-study (one year post-randomization). Range: 0-100; positive values reflect an improvement. Higher values indicate better perceptions of ability to communicate and comprehend.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 105 | 107 | 101
units on a scale | 6.23 (17.38) | 2.97 (14.67) | 3.11 (13.05)

27. Secondary Outcome: Stroke Impact Scale (SIS) Emotion Subscale Score.
Description: Change from baseline to end-of-study (one year post-randomization). Range: 0-100; positive values reflect an improvement. Higher values indicate better perceptions of mood and emotional control.
Time Frame: Baseline to 1 year post-randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care
Number analyzed (Participants) | 105 | 107 | 101
units on a scale | 3.49 (17.81) | 3.63 (17.21) | 3.36 (15.52)

28. Secondary Outcome: Motor Activity Log 28 QOM (MAL-28)
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

29. Secondary Outcome: EQ5D
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

30. Secondary Outcome: Satisfaction With Life Scale (SWLS)
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

31. Secondary Outcome: Single-Item Subjective Quality of Life Measurement (SQOL)
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

32. Secondary Outcome: Reintegration to Normal Living Index (RNLI)
Time Frame: Baseline to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

33. Other Pre Specified Outcome: Monthly Telephone Interviews
Description: A monthly telephone interview with the participant to ascertain information about health status, healthcare utilization, medications, other therapies, and adverse events. Some of these data are reported in the adverse event section. Other data (e.g. those related to healthcare utilization) are part of the secondary analyses presently underway. Until published, these are embargoed information. Once published, these data will be made available via ClinicalTrials.gov.
Time Frame: monthly, beginning 30 days post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

34. Other Pre Specified Outcome: Post-Intervention Interview
Description: A multiple question survey interview, administered by a non-treating, unblinded member of the recruiting team. The participant was asked a set of questions to assess the extent to which critical components of the investigational intervention (e.g. impairment mitigation, session intensity, participant chosen tasks, therapist-participant collaboration) were incorporated into each assigned therapy group. Publication of secondary analyses (outcome measures #5-25) are underway, and until published, they are embargoed information. Once published, these data will be made available via ClinicalTrials.gov.
Time Frame: 16-20 weeks post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

35. Other Pre Specified Outcome: Exit Interview
Description: A multiple question survey interview, administered by a non-treating, unblinded member of the recruiting team. The participant was asked a set of questions regarding activity since the end of the intervention phase. Participants were also asked to report the perceived value of the intervention and study participation. Publication of secondary analyses (outcome measures #5-25) are underway, and until published, they are embargoed information. Once published, these data will be made available via ClinicalTrials.gov.
Time Frame: Post-intervention to 1 year post-randomization
Reporting Status: Not Posted, anticipated posting 2019-07

ADVERSE EVENTS:
Time Frame: From consent to in-person screening (minimum of 5 days post-stroke) up to one year post-randomization (maximum of 471 days post-stroke). Adverse events were not monitored for individuals with medical record screens only.
Description: Participants were monitored for adverse events during all screening, intervention and evaluation sessions. Additionally, participants or their representatives were contacted by phone monthly to assess health status, health care utilization, medication use and occurrence of adverse events. A single event may involve more that one category.
Groups:
- Screened But Not Randomized: Individuals who consented to an in-person screening assessment for eligibility but were never randomized.
Arm/Group | ASAP Accelerated Skill Acquisition Program | DEUCC Dose-Equivalent Usual & Customary Care | UCC Usual & Customary Care | Screened But Not Randomized
Serious Adverse Events (participants affected / at risk) | 37/119 | 36/120 | 32/122 | 4/772
Other Adverse Events (participants affected / at risk) | 67/119 | 69/120 | 55/122 | 1/772
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASAP Accelerated Skill Acquisition Program (N=119) | DEUCC Dose-Equivalent Usual & Customary Care (N=120) | UCC Usual & Customary Care (N=122) | Screened But Not Randomized (N=772)
Death (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Recurrent Stroke or TIA (Nervous system disorders) | 13 (18) | 9 (13) | 7 (9) | 2 (2)
MI or Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 3 (3) | 4 (6) | 0 (0)
New onset of Cardiac Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5) | 6 (6) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inpatient Hospitalization or ER visit >23 hours (General disorders) | 28 (45) | 32 (46) | 28 (48) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Excessive blood pressure response (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) — Of such severity that it required treatment discontinuation for the day
Unexpected/Other (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) — A serious adverse event that involves a condition/circumstance other than those expected and thus other than those pre-identified
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASAP Accelerated Skill Acquisition Program (N=119) | DEUCC Dose-Equivalent Usual & Customary Care (N=120) | UCC Usual & Customary Care (N=122) | Screened But Not Randomized (N=772)
Fall with No Fracture (General disorders) | 41 (67) | 32 (41) | 23 (28) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 6 (6) | 3 (5) | 0 (0)
Open sore or cuts (Skin and subcutaneous tissue disorders) | 8 (10) | 13 (15) | 4 (6) | 0 (0)
Muscle soreness or pain that persists for more than 48 hours (Musculoskeletal and connective tissue disorders) | 29 (53) | 27 (29) | 29 (38) | 0 (0)
Shoulder pain that limits study participation (Musculoskeletal and connective tissue disorders) | 16 (24) | 17 (19) | 20 (27) | 0 (0)
Excessive blood pressure response (Vascular disorders) | 15 (30) | 15 (18) | 3 (4) | 1 (1)
Dizziness/Fainting (General disorders) | 10 (12) | 13 (14) | 9 (10) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Unexpected SAEs (General disorders) | 10 (11) | 12 (12) | 7 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No